CLINICAL TRIAL: NCT01755442
Title: A Phase 1, Double-blind, Randomized, 2-Way Crossover, Placebo-controlled Study to Investigate the Effect of AMG 151 on 24-hour Ambulatory Blood Pressure and Glucose Levels in Subjects With Type 2 Diabetes Mellitus
Brief Title: Investigate Effect of AMG 151 on 24-hour Ambulatory Blood Pressure & Glucose Levels in Type 2 Diabetes Mellitus Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Amgen determined no further need for this study.
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 20120189
Record Dates: First submitted 2012-11-27; First posted 2012-12-24 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2013-04

CONDITIONS: Diabetes Mellitus
Keywords: Ambulatory blood pressure; Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AMG 151 (Active Comparator)
  Interventions: Drug: AMG 151
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Placebo — Eligible subjects will be randomly assigned (1:1) to receive AMG 151 and matching placebo in 1 of 2 sequences over 2 treatment periods.
  Arms: Placebo
Drug: AMG 151 — Eligible subjects will be randomly assigned (1:1) to receive AMG 151 and matching placebo in 1 of 2 sequences over 2 treatment periods.
  Arms: AMG 151

SUMMARY:
This is a phase 1, randomized, double-blind, placebo-controlled, 2-way crossover study to evaluate the effect of AMG 151 on 24-hour ambulatory blood pressure and glucose levels in subjects with type 2 diabetes mellitus who are on a stable regimen of metformin alone, metformin and a dipeptidyl peptidase-4 inhibitor (DPP4), metformin and a thiazolidinedione (TZD), or metformin, a DPP4, and a TZD for a minimum of 3 months prior to randomization.

ELIGIBILITY:
Inclusion Criteria

* Subjects with type 2 diabetes mellitus
* On a stable regimen of metformin alone, metformin and a DPP4, metformin and a TZD, or metformin, a DPP4, and a TZD for a minimum of 3 months prior to randomization
* Body mass indices > 25 and < 45 kg/m2
* Hemoglobin A1c levels ≥ 7.0% and ≤ 11.0% at screening
* Fasting C-peptide levels ≥ 0.2 nmol/L at screening
* Subject with a history of hypertension must be on a stable antihypertensive treatment (s) (type of medication, dose, and regimen) for at least 6 weeks prior to the first dose of investigational product
* Other criteria may apply

Exclusion Criteria

* Subject has type 1 diabetes mellitus or history of type 1 diabetes mellitus
* Subject has had 2 or more emergency room visits or hospitalizations due to poor glucose control in the 6 months prior to screening
* Poorly controlled hypertension defined as diastolic pressure ≥ 95 mmHg or systolic ≥ 155 mmHg (confirmed by a repeat assessment) at screening
* Triglycerides ≥ 400 mg/dL (4.52 mmol/L) at screening
* Use of any known cytochrome P450 (CYP) inducers within 30 days or 5 half-lives (whichever is longer), prior to receiving the first dose of investigational product.
* Use of any known inhibitors of CYP3A4/P-glycoprotein within the 14 days or 5 half lives (whichever is longer) prior to receiving the first dose of investigational product
* Other criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-11; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Mean 24-hour systolic blood pressure | After 14 days of AMG 151 or placebo treatment

SECONDARY OUTCOMES:
Mean 24-hour diastolic blood pressure | After 14 days of AMG 151 or placebo treatment
Mean 24-hour heart rate | After 14 days of AMG 151 or placebo treatment
24-hour concentration time profile of glucose level from continuous glucose monitoring | Day 1 and day 14 of each period
Fasting plasma glucose and fructosamine | After 13 days of AMG 151 or placebo treatment
Plasma glucose 2 hours after time 0 of mixed meal tolerance test | After 13 days of AMG 151 or placebo treatment
4-hour concentration time profile of glucose after the mixed meal tolerance test | After 13 days of AMG 151 or placebo treatment
Safety end points will include the incidence of treatment emergent adverse events. | Up to 2 Months
Serum AMG 151 concentration | Up to 2 Months
Safety end points will include laboratory safety tests. | Up to 2 Months.
Safety end points will include vital signs. | Up to 2 Months
Safety end points will include ECGs. | Up to 2 Months

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- Research Site, San Diego, California, United States

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com